CLINICAL TRIAL: NCT06712069
Title: The Usefulness of Multimodal Intraoperative Neurophysiologic Monitoring During Brain or Spine Surgeries
Brief Title: Evaluating MIONM Effectiveness in Predicting Postoperative Neurological Deficits Using Combined Modalities
Acronym: MIONM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed El Sakka, assistant lecturer of PMR, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0201578; Assistant Lecturer of PMR (Registry Identifier: Ahmed Mosaad Mohamed Arafa Elsakka)
Record Dates: First submitted 2024-11-15; First posted 2024-12-02 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Spine Condition
Keywords: Multimodal IONM, SSEP, MEP, EMG, brain, spine surgery

STUDY DESIGN:
Intervention Model Description: The interventional study in my work , titled "The Usefulness of Multimodal Intraoperative Neurophysiologic Monitoring During Brain or Spine Surgeries," employs a single-group, prospective observational design to evaluate the efficacy of Multimodal Intraoperative Neurophysiologic Monitoring (MIONM) in preventing postoperative neurological deficits. Below are the key elements of the study model:
  Interventional Study Model :
  Design:
  Type: Interventional, Prospective Observational Single Group Assignment: All participants undergo the same intervention using MIONM during their neurosurgical procedures.
  No Control Group: The outcomes of MIONM use are directly compared with expected standards of care based on existing literature
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Multimodal Intraoperative Neurophysiologic Monitoring (MIONM) Arm (Experimental): This arm involves the application of Multimodal Intraoperative Neurophysiologic Monitoring (MIONM) during neurosurgical procedures. Participants in this arm undergo continuous intraoperative monitoring using a combination of:
  Somatosensory Evoked Potentials (SSEP): Monitoring sensory pathway integrity. Motor Evoked Potentials (MEP): Assessing motor pathway functionality. Electromyography (EMG): Detecting nerve irritation and monitoring cranial and limb muscles.
  The intervention is designed to enhance surgical precision by providing real-time feedback to the surgical team, aiming to prevent postoperative neurological deficits and improve patient outcomes. Pre- and postoperative clinical assessments are conducted to evaluate the effectiveness of MIONM.
  Interventions: Device: Multimodal Intraoperative Neurophysiologic Monitoring (MIONM)

INTERVENTIONS:
Device: Multimodal Intraoperative Neurophysiologic Monitoring (MIONM) — Multimodal Intraoperative Neurophysiologic Monitoring (MIONM) is a real-time, device-based intervention used during neurosurgical procedures to monitor and preserve the integrity of neural pathways. It combines the following modalities:
  Somatosensory Evoked Potentials (SSEP): Monitors sensory pathways by stimulating peripheral nerves and recording cortical responses.
  Motor Evoked Potentials (MEP): Assesses motor pathways via transcranial stimulation and muscle response evaluation.
  Electromyography (EMG): Detects nerve irritation and monitors muscle activity during surgery.
  This intervention provides critical real-time feedback to the surgical team, enabling immediate adjustments to prevent neurological damage and enhance surgical outcomes. The Cascade IOMAX system is the primary device used in this study for implementing MIONM.

SUMMARY:
Objective: This study aimed to integrate findings from spinal and cranial surgeries with existing literature, emphasizing the role of Intraoperative Neurophysiological Monitoring (IONM) in improving surgical outcomes through best practices.

Methodology: Multimodal IONM, including motor evoked potential (MEP), somatosensory evoked potential (SSEP), and electromyography (EMG), was utilized in surgeries at Duke University Hospitals. Challenges included a small sample size and limited access to medical records.

Findings:

Effectiveness of IONM: High sensitivity (97.73%), specificity (83.33%), and predictive value of multimodal IONM confirmed its role in detecting intraoperative neurological injuries and optimizing outcomes.

Demographics: Analysis of 50 cases (58% male, aged 13-67 years) revealed demographic influences on surgical challenges and outcomes.

IONM Alerts: A 50% reduction in MEP/SSEP amplitudes was a critical criterion, with reversible alerts accounting for 70%, emphasizing the dynamic nature of neural responses.

Alert Causes & Management: Excessive dissection was a common cause of alerts. Interventions like warm saline irrigation and surgical pauses mitigated risks.

Outcome Associations: Most patients (88%) experienced no new postoperative deficits, with significant associations between alert reversibility and deficit occurrence.

Statistical Insights:

Predictive Value: Strong correlations were observed between alert patterns and postoperative outcomes, with SSEP/MEP alerts reliably predicting neurological deficits.

Technology & Resources: Modern devices, updated technology, and skilled staff were critical for high-quality results, highlighting the adage that "poor monitoring is worse than no monitoring."

Contextual Observations:

Heterogeneity of Cases: Diagnoses ranged from cervical intramedullary tumors to lumbar canal stenosis, requiring tailored interventions.

EMG Utility: EMG showed stability with fewer alerts, proving beneficial in specific surgeries.

Corrective Measures: Adjustments in mean arterial blood pressure and steroid use showcased adaptive intraoperative strategies.

Protocol Gaps: The absence of standardized IONM alert response protocols was noted, underscoring the need for future research.

DETAILED DESCRIPTION:
Detailed Description:

The discussion emphasizes the importance of intraoperative neurophysiological monitoring (IONM) in enhancing surgical safety during spinal and cranial procedures. Multimodal IONM (MIONM), incorporating somatosensory evoked potentials (SSEP), motor evoked potentials (MEP), and electromyography (EMG), serves as a critical tool for real-time neurological monitoring during these complex operations.

MIONM is highlighted for its ability to detect intraoperative neurological changes, enabling timely interventions. Factors such as patient demographics and case heterogeneity, including diverse diagnoses like craniotomy, lumbar canal stenosis, scoliosis, and cervical intramedullary tumors, underscore the need for tailored surgical approaches. The integration of modern equipment and experienced personnel ensures the delivery of high-quality monitoring results.

The discussion also explores the challenges in managing IONM alerts, including causes like over-dissection, hypoperfusion, and excessive cord manipulation. A multimodal approach to handling alerts includes interventions such as positional adjustments, warm saline irrigation, and optimizing blood flow. The absence of standardized protocols for responding to alerts highlights the need for future research to develop evidence-based guidelines.

Further research is encouraged to refine IONM methodologies, customize surgical strategies based on patient-specific factors, and establish standardized alert response protocols to optimize outcomes in spinal and cranial surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 12 years.
2. Various brain or spinal pathologies that are indicated for (IONM) such as (cerebellopontine angle tumors, scoliosis, epidural abscesses, arteriovenous malformations, canal stenosis, tumor resection, and craniotomies.
3. Medically fit for surgery.

Exclusion Criteria:

1. Unobtainable or poor baselines (both MEPs and SSEPs).
2. Patients with a motor power grade of 1 or below.
3. Presence of vascular clips, intracranial electrodes, pacemakers, other implanted biomechanical equipment, cortical lesions, skull defects, increased intracranial pressure, and history of epilepsy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
rate of occurrence of New Postoperative Neurological Deficits | Evaluated within one-week post-surgery.
  The primary outcome is the proportion of patients who develop new neurological deficits (motor, sensory, or combined) after undergoing neurosurgical procedures with Multimodal Intraoperative Neurophysiologic Monitoring (MIONM). These deficits will be assessed through detailed clinical examinations pre- and post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Imam, Phd in PMR, Study Chair — Alexandria University , Faculty of Medicine
Locations (1):
- Alexandria Main University Hospital (AMUH), Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared with other researchers to protect participant confidentiality and privacy. Additionally, institutional and ethical guidelines restrict the sharing of such data outside the scope of this study. The collected data will be used solely for the analysis and reporting of study results

REFERENCES:
- [Background] 1. Brandmeier S, Taskiran E, Bolukbasi FH, Sari R, Elmaci I. Multimodal intraoperative neurophysiological monitoring in neurosurgical oncology. Turk Neurosurg 2018;28(2):204-10. 2. Novak K, Oberndorfer S. Electrophysiology and intraoperative neurophysiological monitoring. In: Handbook of Clinical Neurology 2012; 104:149-61. 3. Miró Lladó J, López-Ojeda P, Pedro J, Marnov A, Contreras L, Pariente L, et al. Evaluation of multimodal intraoperative neurophysiologic monitoring during supratentorial aneurysm surgery: a comparative study. Neurosurg Rev 2022 ;45(3):2161-73. 4. Tsirikos AI, Duckworth AD, Henderson LE, Michaelson C. Multimodal intraoperative spinal cord monitoring during spinal deformity surgery: efficacy, diagnostic characteristics, and algorithm development. Med Princ Pract 2020;29(1):6-17. 5. Cavinato M, Vittoria F, Piccione F, Masiero S, Carbone M. The value of intraoperative neurophysiological monitoring during positioning in pediatric scoliosis correction: A case report. Clin Neurophysiol Pract 2022; 7:366-71. 6. Park JH, Hyun SJ. Intraoperative neurophysiological monitoring in spinal surgery. World J Clin Cases 2015;3(9):765.

DOCUMENTS (3):
  • Study Protocol (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT06712069/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT06712069/SAP_001.pdf
  • Informed Consent Form (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT06712069/ICF_002.pdf